CLINICAL TRIAL: NCT05650437
Title: Impact of Ultraviolet Radiation on Bone Density and Muscle Strength in Postmenopausal Women: A Randomized Controlled Study
Brief Title: Impact of Ultraviolet Radiation on Bone Density and Muscle Strength in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 66
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultraviolet therapy group (Active Comparator): 35 women will undergo three weekly sessions of UV therapy in addition to routine aerobic activity and vitamin D supplements (800 IU) daily for three months
  Interventions: Device: Ultraviolet Radiation; Behavioral: Aerobic exercise; Dietary Supplement: Vitamin D supplementation
- Non Ultraviolet therapy group (Active Comparator): 35 women will undergo three weekly sessions of routine aerobic activity and vitamin D supplements (800 IU) daily for three months
  Interventions: Behavioral: Aerobic exercise; Dietary Supplement: Vitamin D supplementation

INTERVENTIONS:
Device: Ultraviolet Radiation — The therapist cut three holes, each measuring 2 by 2 cm, into a piece of cardboard that was about 4 by 20 cm in size.The first hole was exposed for 90 seconds, the second for 60 seconds, and the third for 30 seconds
  Arms: Ultraviolet therapy group
Behavioral: Aerobic exercise — The postmenopausal women in groups (A and B) exercised on the treadmill; women should always warm up before beginning exercise and stop if they experience pain or shortness of breath. Each session lasted 30 minutes and included 5 minutes of warming up and 20 minutes of walking at 60% of their maximum heart rate (MHR). The maximum heart rate that the circulatory system can support during physical exercise is MHR=220. Three sessions a week for three months, followed by a five-minute cool-down
Dietary Supplement: Vitamin D supplementation — Throughout three months, vitamin D supplements (800 IU) will be given to all postmenopausal women in both groups (A&B)

SUMMARY:
70 postmenopausal women, aged 50 to 60, who are vitamin D deficient and diagnosed with osteoporosis or osteopenia with T score of DEXA of lumbar spine (L1 to L4) was less than or equal -1 and their body mass index between 25 and 30 kg/m2. They will be divided into two groups by randomization. 35 postmenopausal women in Group (A) will undergo three weekly sessions of UV therapy in addition to routine aerobic activity and vitamin D supplements (800 IU) daily for three months. For three months, group (B), which consists of 35 postmenopausal women, will undergo daily aerobic exercise and vitamin D supplementation (800 IU) only.

The amount of serum 25-hydroxyvitamin D was measured using ELISA kits, bone mineral density of lumber spine was measured by dual energy X-ray absorptiometry (DEXA), and the torque of knee flexors and extensors was evaluated using the Biodex System 3 isokinetic dynamometer,

DETAILED DESCRIPTION:
Group (A): This group covers a sum of 35 postmenopausal women who underwent three weekly sessions of UV light therapy in addition to daily vitamin D supplements of 800 IU.

Ultraviolet therapy device It was an ultraviolet arc lamp made of a low-pressure mercury discharge tube with an internal phosphor coating. The chemical makeup of the phosphor utilized determined the specific wavelength and output of each light (mixtures of phosphates, borates, and silicates). This produces a sizable amount of UVA and UVB but none of UVC. The spectrum of the radiation: is 280-320 nm. Postmenopausal women in the group received treatment with quartz of the type 4004/2n- Verret (A).

Using dose-response assessment, which is graded according to the individual's erythema response and is classified as E1, Second-degree erythema (E2), Third-degree erythema (E3), and Fourth-degree erythema, the physical therapist determined the postmenopausal woman's sensitivity to UV before applying UV (E4).

The physical therapist instructed each case to wear safety glasses (goggles) to protect her eyes from UV, and treatment duration was calculated as a percentage of the MED of UV. The woman was then instructed to take off all of her clothes and wash her abdomen. After describing the steps to the woman and requesting that she avoid looking at the bulb due to the risk of eye damage. The therapist cut three holes, each measuring 2 by 2 cm, into a piece of cardboard that was about 4 by 20 cm in size.

Subsequently, the region around the cardboard was covered with a cloth to prevent the skin nearby from being exposed to radiation by placing the cardboard on the abdomen. The lamp was turned on and positioned 70 cm away and perpendicular to the abdominal region. Before turning toward the woman, the arc lamp needed five to ten minutes to warm up and attain maximum power. The UV beam was pointed straight at the abdomen region after the lamp had achieved maximum power, which activated the timer. The three holes were exposed to UV light for 30 seconds at a time, after which two holes were covered and one was left unattended for the following 30 seconds.

The first hole was exposed for 90 seconds, the second for 60 seconds, and the third for 30 seconds by this protocol. Then, instruct the woman to document the region's reaction for 24 hours after exposure. The area that experienced minor skin reddening within eight hours and faded within twenty-four hours was given MED treatment. The minimum erythemal dose (MED) or E1 was the desired dose in this study.

Following the determination of the MED for each woman, the UV session was conducted as follows: To maximize exposure of the portion being treated and prevent unnecessary exposure of other parts, the postmenopausal lady was directed to remove clothing from the lower abdomen and lie in a supine position.

As for the rest of the body, which did not require exposure, it was covered. Goggles are necessary to shield the eyes from exposure. After that, the ultraviolet Arc lamp was adjusted so that it is positioned approximately 70 cm above the lower abdominal region in a perpendicular position. By the MED for each lady that was spotted, the lamp was switched on and the timer was changed.

The lamp was turned off and moved away from the postmenopausal woman by the end of the therapy period. Any noticeable reaction to the therapy was recorded within the three treatment sessions per week which were administered for a total of three months.

Aerobic exercise The postmenopausal women in groups (A and B) exercised on the treadmill; women should always warm up before beginning exercise and stop if they experience pain or shortness of breath. Each session lasted 30 minutes and included 5 minutes of warming up and 20 minutes of walking at 60% of their maximum heart rate (MHR). The maximum heart rate that the circulatory system can support during physical exercise is MHR=220. Three sessions a week for three months, followed by a five-minute cool-down [10].

Vitamin D supplementation Throughout three months, vitamin D supplements (800 IU) were given to all postmenopausal women in both groups (A&B).

The Group (B): This group comprises of 17 postmenopausal women who completed 3 months of daily aerobic exercise and vitamin D supplementation (800 IU).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women who did not engage in any recreational physical activity in the previous three months Low bone mineral density (BMD) at their spine and/or femoral neck met the inclusion criteria.

They are in good health. body mass index (BMI) ranged from 25 to 30 kg/m2, ages ranged from 50 to 60

Exclusion Criteria:

* mental, neurological, Vestibular, cardiovascular, metabolic disease, musculoskeletal disorders with lower limb deformity, visual or hearing impairment undergone hormone replacement therapy. any medication that affected their balance or photosensitizing medications like aspirin, tetracycline, and Chlorothiazide

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
T-score of mineral density of lumber spine | 3 months from treatment
  measured by dual energy X-ray absorptiometry
Peak Torque of knee flexors and extensors | 3 months from treatment
  The isokinetic dynamometer for the Biodex System 3, Biodex Medical System, Shirley, New York, USA, was recommended to be used in the current study [11]. It was adopted in the study to evaluate the muscular strength of the knee flexors and extensors in all postmenopausal women in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Maged, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No